CLINICAL TRIAL: NCT04340999
Title: Electrophysiological Evaluation of Motor Dysfunction in Liver Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Reem Mahmoud Mohamed Ali Gabr, Resident of Clinical neurophysiology- Kasr alainy-Cairo University, Kasr El Aini Hospital
Other Study IDs: Electrophysiology - cirrhosis
Record Dates: First submitted 2020-04-04; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Liver Cirrhoses; Peripheral Neuropathy
Keywords: Liver cirrhotic patients- Motor Dysfunction-Fatigue.
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Manifested Group: Manifested Group , enrolled patients who had any of the following manifestations(Fatigue,muscle cramps or numbness)
  Interventions: Diagnostic Test: Nerve conduction studies and Quantitative EMG ( MUNE and IPA)
- Non-Manifested Group: Non-manifested group in which enrolled patients didn't report any of the following manifestations
  Interventions: Diagnostic Test: Nerve conduction studies and Quantitative EMG ( MUNE and IPA)

INTERVENTIONS:
Diagnostic Test: Nerve conduction studies and Quantitative EMG ( MUNE and IPA) — Nerve Conduction Studies: Electrophysiological method that tests the presence/absence of peripheral neuropathy.
  MUNE: Electrophysiological technique that assess number of motor units. IPA: Electrophysiological method that assess interference pattern and hence, borderline cases of neuropathy/ myopathy

SUMMARY:
cross sectional observational study, aimed to assess the electrophysiological function of the motor units in liver cirrhotic patients.

DETAILED DESCRIPTION:
Liver cirrhosis is a global health problem which could be associated with several neurological manifestations. The associated peripheral neuropathy could be assessed by conventional nerve conduction studies.

Objective: The study aims at early detection of peripheral neuropathy among patients of liver cirrhosis by conventional nerve conduction studies and quantitative EMG methods. In addition, the study aims at finding out correlation between peripheral neuropathy and severity of the liver cirrhosis.

Methods: This a cross-sectional study conducted on fifty-six liver cirrhotic patients, that had been recruited from the Endemic medicine department/outpatient clinics and their age-gender matched sixty-one healthy controls. The recruited patients were clinically assessed .Both conventional nerve conduction studies and quantitative EMG techniques in the form of MUNE calculation, using modified spike -triggered technique and IPA ratio evaluation were performed for the allocated cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age interval range between 18 and 60 years (To avoid maturational changes and aging process on motor unit number).
* Liver cirrhotic patients( including compensated and decompensated patients);

  * Presenting hematemesis/melena and/or ascites.
  * Diagnosis of liver cirrhosis is confirmed by abdominal ultrasound

Exclusion Criteria:

* Patients with identifiable cause of peripheral neuropathy (e.g. diabetic patients) .
* Patients who developed hepatocellular carcinoma (to avoid para-neoplastic syndrome e.g. peripheral neuropathy)
* Patients with other non-hepatic chronic illness such as: patients with renal disease (to avoid other causes of metabolic neuropathies).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifty-Six liver cirrhotic patients that were recruited from the Endemic medicine department and its outpatient clinics, at Kasr Alainy hospitals, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Early detection of peripheral neuropathy among liver cirrhotic patients. | baseline
  * Using nerve conduction studies of the: left ulnar,left posterior tibial and right deep peroneal motor nerves;assess their distal latency (measured in milliseconds) ,amplitude (measured in millivolts) and conduction velocities (measured in m/s).In addition , to sensory studies of the left ulnar and right sural sensory nerves; assessment of peak latency (measured in milliseconds) , amplitude (measured in microvolts) and their conduction velocities(measured in m/s) .
  * Compare the values with our normative values.
  * Detect evidence of peripheral neuropathy ( increased in distal latency above the upper limit of its normal value, decreased conduction velocity below the lower limit of its normal value and decreased amplitude below lower limit of its normal value).
  * A minimum of three variables in two or more nerves are required to diagnose polyneuropathy as referenced by (Meulstee & Van Der Meche , 1995).

SECONDARY OUTCOMES:
Detection of correlation between neuropathy and severity of liver cirrhosis. | baseline
  Finding out any correlation between peripheral neuropathy and severity of liver cirrhosis:
  * Comparing between patients with evidence of peripheral neuropathy (as detected by nerve conduction studies) and those without evidence of peripheral neuropathy versus the severity of their liver disease ( as assessed by Child-Pugh class) using Mann Whitney U test; to find out if their is statistical difference between them or not; denoting the presence/absence of correlation between peripheral neuropathy and the severity of the liver disease.
Motor unit number estimation using Spike-Triggered method. | Baseline
  * Estimation of motor unit number using Spike-Triggered method in liver cirrhotic patients and age/gender healthy controls to find out of there is statistical difference between them.
  * Decline in MUNE values denotes loss of motor neurons.
Correlation of MUNE values to fatigue | Baseline
  * Comparing between liver cirrhotic patients who reported fatigue(as part of their neurological symptoms) versus those who didn't report fatigue, regarding their MUNE values; using Mann Whitney U test.
  * If there is statistical difference between them; there would be correlation between loss of motor units and fatigue reported by the patients(this assumption was based on (Heckman & Enoka, 2012) &(Mota et al., 2020) conclusions that there is positive correlation between fatigability and loss of motor units.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Teaching Hospital-Clinical Neurophysiology Unit, Giza, Egypt

REFERENCES:
- [Background] • Abdel-Razek, W., Hassany, M., Kabil, K., Ammar, I., Dabous, H., Doss, W., ... & El-Serafy, M. (2019). The World's Largest Hepatitis C Screening Program in Egypt. Journal of Hepatology (Vol. 70, pp. 144-145). • Abrams, G. A., Concato, J., & Fallon, M. B. (1996). Muscle cramps in patients with cirrhosis. American Journal of Gastroenterology, 91(7). • Aggarwal A, Nicholson G. (2002).Detection of preclinical motor neurone loss in SOD1 mutation carriers using motor unit number estimation. Journal of Neurology, Neurosurgery & Psychiatry; 73(2):199-201. • Amodio, P., & Gatta, A. (2005). Neurophysiological investigation of hepatic encephalopathy. Metabolic brain disease, 20(4), 369-379. • Arabadzhiev, T. I., Dimitrov, G. V., Dimitrov, A. G., Chakarov, V. E., & Dimitrova, N. A. (2008). Factors affecting the turns analysis of the interference EMG signal. Biomedical Signal Processing and Control, 3(2), 145-153. • Barkhaus, P. E. (2001). Motor Unit Action Potential Quantitation. In An AAEM workshop. Rochester, Minn: American Association of Electrodiagnostic Medicine (Vol. 2). • Bessou, P., Emonet-Dénand, F., & Laporte, Y. (1965). Motor fibres innervating extrafusal and intrafusal muscle fibres in the cat. The Journal of Physiology, 180(3), 649-672. • Blok, J. H., van Dijk, J. P., Drost, G., Zwarts, M. J., & Stegeman, D. F. (2002). A high-density multichannel surface electromyography system for the characterization of single motor units. Review of Scientific Instruments, 73(4), 1887-1897.